CLINICAL TRIAL: NCT02753101
Title: Biodistribution and Pharmacokinetic Determination of the PET Radiopharmaceutical [18F]FTC-146 Using PET/MRI in Healthy (Asymptomatic) Volunteers and in Patients With CRPS and Sciatica
Brief Title: [18F]FTC-146 PET/MRI in Healthy Volunteers and in CRPS and Sciatica
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Sandip Biswal, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 32231
Record Dates: First submitted 2016-04-22; First posted 2016-04-27 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Complex Regional Pain Syndrome; Sciatica
Keywords: Positron Emission Tomography; Magnetic Resonance Imaging; PET/MRI; sigma-1 receptor; radiopharmaceutical; complex regional pain syndrome; sciatica; chronic pain
MeSH Terms: conditions — Complex Regional Pain Syndromes; Sciatica; Chronic Pain | interventions — 6-(3-fluoropropyl)-3-(2-(azepan-1-yl)ethyl)benzo(d)thiazol-2(3H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): [18F]-FTC-146
  Interventions: Drug: [18F]-FTC-146

INTERVENTIONS:
Drug: [18F]-FTC-146 — 10 mCi± 1 mCi of [18F]FTC-146 intravenously
  Other Names: Sigma-1 receptor radioligand

SUMMARY:
Chronic pain can result from injured or inflamed nerves, as occurs in people suffering from sciatica and CRPS. These nerve injuries or regions of nerve irritation are often the cause of pain in these conditions, but the current diagnostic tools are limited in pinpointing the area of origin. Several studies have implicated involvement of sigma-1 receptors in the generation and perpetuation of chronic pain conditions, others are investigating anti sigma-1 receptor drugs for the treatment of chronic pain. Using the sigma-1 receptor (S1R) detector and experimental radiotracer [18F]FTC-146 and positron emission tomography/magnetic resonance imaging (PET/MRI) scanner, the researchers may potentially identify the source of pain generation in patients suffering from complex regional pain syndrome (CRPS) and chronic sciatica. The ultimate goal is to assist in the optimization of pain treatment regimens using an [18F]FTC-146 PET/MRI scan.

The study is not designed to induce any physiological/pharmacological effect.

DETAILED DESCRIPTION:
Participants are either pain free (control) or will be recruited based on established criteria for sciatica or CRPS. A signed consent will be obtained from willing participants.

For the PET/MRI scan, the participants will be injected with [18F]FTC-146 intravenously. After injection, simultaneous PET and MRI scans will be acquired using a hybrid PET/MRI scanner. Throughout scanning, participants will be monitored for blood pressure, temperature, heart rate and pulse oximetry. Participants will be asked to void their bladder as frequently as they can to reduce radiation exposure. Following the scan, participants will be contacted to check for adverse drug events, and any events will be recorded in the case report.

Evidence in the literature points strongly toward an involvement of S1 receptors in nervous system inflammation, which is known to be an important biologic disease/disorder mechanism for maintenance and perpetuation of chronic pain.

The main purpose of this research study is to image and identify activated pain pathways in human subjects using [18F]FTC-146 PET/MRI.

ELIGIBILITY:
Inclusion Criteria:

General:

* At least 18 years of age
* Either male or female

Sciatica:

* History of pain shooting down a leg below the knee, to the foot or toes
* Visual analog scale (VAS) at enrollment of >4 with leg pain greater in intensity than the back pain
* Focal disc herniation on MRI correlating with radicular symptoms defined as pain or paresthesias into the leg.
* Examination with correlating radicular signs defined as any of the following:
* pain reproduction with straight-leg-raising (pain shooting down the leg with less than 60 degrees elevation)
* radicular pattern sensory changes (such as numbness or paresthesias) in the same area as pain
* signs of radiculopathy (weakened hallux extension and/or Achilles tendon reflex)
* The above inclusion criteria can be met OR individuals who have been determined to have a very high clinical suspicion of having Sciatica as determined by the referring pain specialist can be included. This suspicion will be documented in the patient's medical record.

CRPS:

* Disease duration of 6 months or longer
* Continuing pain, which is disproportionate to any inciting event
* Must report at least one symptom in three of the four following categories:

  1. Sensory: Reports of hyperesthesia and/or allodynia
  2. Vasomotor: Reports of temperature asymmetry and/or skin color changes and/or skin color asymmetry
  3. Sudomotor/Edema: Reports of edema and/or sweating changes and/or sweating asymmetry
  4. Motor/Trophic: Reports of decreased range of motion and/or motor dysfunction (weakness, tremor, dystonia) and/or trophic changes (hair, nail, skin)
* Must display at least one sign at time of evaluation In two or more of the following categories:

  1. Sensory: Evidence of hyperalgesia (to pinprick) and/or allodynia (to light touch and/or temperature sensation and/or deep somatic pressure and/or joint movement)
  2. Vasomotor: Evidence of temperature asymmetry ( >1°C) and/or skin color changes and/or asymmetry
  3. Sudomotor/Edema: Evidence of edema and/or sweating changes and/or sweating asymmetry
  4. Motor/Trophic: Evidence of decreased range of motion and/or motor dysfunction (weakness, tremor, dystonia) and/or trophic changes (hair, nail, skin)
* There is no other diagnosis that better explains the signs and symptoms
* For research purposes, diagnostic decision rule will be at least one symptom in all four symptom categories and at least one sign (observed at evaluation) in two or more sign categories.
* The above inclusion criteria can be met OR individuals who have been determined to have a very high clinical suspicion of having CRPS as determined by the referring pain specialist can be included. This suspicion will be documented in the patient's medical record.

Exclusion Criteria:

General:

* Another active disorder which could explain the symptoms in the opinions of the investigator
* Failure to give informed consent
* Presence of MRI-incompatible materials/devices
* Any medication that may affect pain or 18F-FTC-146 uptake or adverse drug interactions with steroids or amino amide local anesthetics (e.g. lidocaine, bupivacaine, ropivacaine)
* Pregnant or nursing
* Ongoing menstrual period
* Severe comorbid conditions
* Unable to read or complete questionnaires in English
* Any other condition, which in the opinion of the investigator would impede compliance or hinder completion of the study

Sciatica:

* Any condition that may interfere with interpretation of 18F-FTC-146 uptake in the region of the pelvis, thighs or lower spine including, but not limited to,

  1. Spinal, hip or pelvic surgery or prosthesis
  2. Cancer
  3. Radiation therapy
  4. Autoimmune disorders
  5. Current infections
  6. Inability to void bladder completely, such as in prostatic enlargement
  7. Any urinary retention, such as in outlet obstruction, hydronephrosis etc.
  8. Cauda equina syndrome
  9. Developmental spinal deformities
  10. Scoliosis >20 degrees
  11. Spondylolysis
  12. Vertebral fractures
  13. Inflammatory spondylopathy
  14. Prior lumbar surgery

      CRPS:
* Presence of current or past pulmonary, hepatic, renal disease, arthritis, hematopoietic, and neurological diseases not related to CRPS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-16 (Actual)

PRIMARY OUTCOMES:
Biodistribution of [18F]FTC-146 | an estimated average of 2 hours
  Biodistribution of [18F]FTC-146 will be analyzed by drawing regions of interest (ROI) for the reported organs on the PET/MRI images. Processing software will quantify the amount of [18F]FTC-146 uptake within the ROI's and display the amount in terms of standardized uptake values (SUV's).
  Biodistribution data will be obtained by drawing regions of interest (ROI's) around organs on the PET/MRI images. Processing software will quantify the amount of [18F]FTC-146 uptake within the ROI's and display the amount in terms of standardized uptake values (SUV's).
  Pharmacokinetic data will be calculated using kinetic analysis (mathematical modeling) of [18F]FTC-146 clearance from the blood.

SECONDARY OUTCOMES:
Dosimetry of [18F]FTC-146 | an estimated average of 2 hours
  Dosimetry calculations will be determined using the biodistribution (reported as a primary outcome measure) and pharmacokinetics of the tracer in human organs.
Incidence of Adverse Events | Baseline and up to 7 days after tracer injection
  [18F]FTC-146 Single IV Treatment-Emergent Adverse Events will be established by collectively assessing real-time vitals monitoring during scans, serial clinical lab work (i.e. blood tests), and patient symptomatic report at baseline and up to 7 days post-injection.

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Biswal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Background] James ML, Shen B, Nielsen CH, Behera D, Buckmaster CL, Mesangeau C, Zavaleta C, Vuppala PK, Jamalapuram S, Avery BA, Lyons DM, McCurdy CR, Biswal S, Gambhir SS, Chin FT. Evaluation of sigma-1 receptor radioligand 18F-FTC-146 in rats and squirrel monkeys using PET. J Nucl Med. 2014 Jan;55(1):147-53. doi: 10.2967/jnumed.113.120261. Epub 2013 Dec 12. PMID 24337599
- [Background] James ML, Shen B, Zavaleta CL, Nielsen CH, Mesangeau C, Vuppala PK, Chan C, Avery BA, Fishback JA, Matsumoto RR, Gambhir SS, McCurdy CR, Chin FT. New positron emission tomography (PET) radioligand for imaging sigma-1 receptors in living subjects. J Med Chem. 2012 Oct 11;55(19):8272-8282. doi: 10.1021/jm300371c. Epub 2012 Sep 20. PMID 22853801
- [Background] Fletcher JW, Djulbegovic B, Soares HP, Siegel BA, Lowe VJ, Lyman GH, Coleman RE, Wahl R, Paschold JC, Avril N, Einhorn LH, Suh WW, Samson D, Delbeke D, Gorman M, Shields AF. Recommendations on the use of 18F-FDG PET in oncology. J Nucl Med. 2008 Mar;49(3):480-508. doi: 10.2967/jnumed.107.047787. Epub 2008 Feb 20. PMID 18287273
- [Background] Puente B, Nadal X, Portillo-Salido E, Sanchez-Arroyos R, Ovalle S, Palacios G, Muro A, Romero L, Entrena JM, Baeyens JM, Lopez-Garcia JA, Maldonado R, Zamanillo D, Vela JM. Sigma-1 receptors regulate activity-induced spinal sensitization and neuropathic pain after peripheral nerve injury. Pain. 2009 Oct;145(3):294-303. doi: 10.1016/j.pain.2009.05.013. Epub 2009 Jun 7. PMID 19505761
- [Background] Entrena JM, Cobos EJ, Nieto FR, Cendan CM, Gris G, Del Pozo E, Zamanillo D, Baeyens JM. Sigma-1 receptors are essential for capsaicin-induced mechanical hypersensitivity: studies with selective sigma-1 ligands and sigma-1 knockout mice. Pain. 2009 Jun;143(3):252-261. doi: 10.1016/j.pain.2009.03.011. Epub 2009 Apr 17. PMID 19375855
- [Background] Maurer AH. Combined imaging modalities: PET/CT and SPECT/CT. Health Phys. 2008 Nov;95(5):571-6. doi: 10.1097/01.HP.0000334064.46217.20. PMID 18849691